CLINICAL TRIAL: NCT02954549
Title: Genomics of Vitamin D Supplementation and Warfighter Nutritional Resilience
Brief Title: Vitamin D Supplementation in Warfighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: TriService Nursing Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HU001-15-1-TS05
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Vitamin D Deficiency Disease
Keywords: vitamin D deficiency, genomics, vitamin D supplementation
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy control group (Active Comparator): Subjects in this arm have a normal serum level of 25(OH)D, >30 ng/mL. Subjects submit to blood draws and biometric tests (DXA, body composition, BP) and questionnaires on 3 occasions. They do not receive vitamin D3 supplementation.
  Interventions: Dietary Supplement: Vitamin D3
- Low dose supplementation group (Experimental): Subjects in this group have been identified as having a level of 25(OH)D of < 30 ng/mL and are randomized to receive vitamin D3 supplementation of 2000 IU daily for 3 months.
  Interventions: Dietary Supplement: Vitamin D3
- High dose supplementation group (Experimental): Subjects in this group have been identified as having a level of 25(OH)D of <30 ng/mL and are randomized to receive vitamin D3 supplementation of 5000 IU daily for 3 months.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — As in Arms
  Other Names: Cholecalciferol

SUMMARY:
A genomics-based approach will target specific genes that may explain the response in biomarkers and symptoms before and after supplementation. One objective is to generate evidence-based recommendations for vitamin D supplementation in Soldiers who often experience musculoskeletal disorders and immune dysfunction impacting physical performance and military readiness. The investigation is designed to address these specific aims: 1) explore vitamin D status in 105 Service Members to determine common symptoms associated with deficiency; 2) examine the effect of vitamin D levels on gene expression from select genes known to influence metabolism, bone density, and immune function; and 3) evaluate changes in gene expression between groups receiving high or low supplementation, and compare to healthy controls. Follow-up at 15 months will evaluate circulating vitamin D.

DETAILED DESCRIPTION:
A genomics-based approach will target identified candidate genes and search for variants that may explain the response observed in biomarkers and symptoms when deficient individuals are repleted. The long-term objective of this study is to translate findings from next-generation sequencing (NGS) technology into clinically meaningful data regarding vitamin D supplementation for Service Members (SM) who may be at risk for musculoskeletal disorders and immune dysfunction that impacts physical performance and military readiness. We propose the following specific aims: 1) explore the phenotypic expression of vitamin D status in a cohort of SM to determine common symptoms associated with deficiency/insufficiency states; 2) examine the effect of vitamin D levels on broad gene expression from carefully chosen candidate genes known to influence vitamin D status, bone density, and immune function; 3) evaluate changes in gene expression levels between and within groups supplemented with low vs high vitamin D, and compare to healthy controls, and 4) examine the relationship between vitamin D deficiency and the clinically relevant outcomes of stress fracture and high blood pressure before and after supplementation to a therapeutic plasma level of 25(OH)D. This prospective, randomized, double-blind trial will enroll 105 SM in the Northwest to evaluate frequency, symptoms, and genomic expression of vitamin D levels using survey instruments, immunologic and bone biomarkers, and NGS of white blood cells pre- and post-supplementation with oral vitamin D over 3 months. Participant follow-up at 12 months will evaluate maintenance of adequate circulating vitamin D; this timeframe represents a typical deployment period.

ELIGIBILITY:
Inclusion Criteria:

- active duty service member, age 18 years or older, ability to read and understand English, not deploying in the next 15 months, and subjectively in good health.

Exclusion Criteria:

- family members, beneficiaries, or civilians, pregnant or currently breastfeeding females, anyone with chronic health problems (e.g. eating disorders, kidney disease, liver disease, intestinal malabsorption), any active duty SM taking >400 IU/day vitamin D supplementation and unwilling to discontinue this, current or healing stress fractures, taking medications for an endocrine disorder, such as synthroid, or those identified as having a high potential for interaction with vitamin D including anti-seizure medications, cyclosporine, and indinavir (Crixivan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
25(OH)D | 15 months
  Serum measure of 25(OH) at baseline, 3 months, and 15 months

SECONDARY OUTCOMES:
Vitamin D gene expression | 3 months
  Gene expression analysis will be used to determine relationship between low and high dose vitamin D supplementation and 25(OH)D levels, blood pressure, bone density, and body fat

CONTACTS AND LOCATIONS:
Overall Officials: Mary S McCarthy, PhD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiscella K, Franks P. Vitamin D, race, and cardiovascular mortality: findings from a national US sample. Ann Fam Med. 2010 Jan-Feb;8(1):11-8. doi: 10.1370/afm.1035. PMID 20065273
- [Background] Yanovich R, Friedman E, Milgrom R, Oberman B, Freedman L, Moran DS. Candidate gene analysis in israeli soldiers with stress fractures. J Sports Sci Med. 2012 Mar 1;11(1):147-55. eCollection 2012. PMID 24149131
- [Background] Carlberg C. Genome-wide (over)view on the actions of vitamin D. Front Physiol. 2014 Apr 29;5:167. doi: 10.3389/fphys.2014.00167. eCollection 2014. PMID 24808867
- [Result] Hossein-nezhad A, Spira A, Holick MF. Influence of vitamin D status and vitamin D3 supplementation on genome wide expression of white blood cells: a randomized double-blind clinical trial. PLoS One. 2013;8(3):e58725. doi: 10.1371/journal.pone.0058725. Epub 2013 Mar 20. PMID 23527013